CLINICAL TRIAL: NCT05582122
Title: SURVEILLE-HPV: National, Multicenter, Open-label, Randomized, Phase II Study Evaluating HPV16 Circulating DNA as Biomarker to Detect the Recurrence, in Order to Improve Post Therapeutic Surveillance of HPV16-driven Oropharyngeal Cancers
Brief Title: SURVEILLE-HPV: Evaluation of HPV16 Circulating DNA as Biomarker to Detect the Recurrence, in Order to Improve Post Therapeutic Surveillance of HPV16-driven Oropharyngeal Cancers
Acronym: SURVEILLE-HPV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UC-HNG-2209
Record Dates: First submitted 2022-10-11; First posted 2022-10-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Oropharynx Squamous Cell Carcinoma
Keywords: HPV16; CtDNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard follow-up monitoring (16 visits over 5 years) (No Intervention): Patients enrolled in the control arm will be monitored according to SFORL guidelines. Physical Examination (PE) will be carried out:
  - every 2 months the 1st year, every 3 months the 2nd year, every 4 months the 3rd year, every 6 months at 4 and 5 years.
  Annual chest CT scan will be performed for current smokers & for those who have quit smoking less than 15 years ago.
- Lightened follow-up visits frequency (9 visits over 5 years), with HPV16 Ct-DNA dosing (Experimental): Physical Examinations (with HPV16 Ct-DNA dosing) planned at Months 4,8,12,18,24,30,36,48,60 post treatment.
  Annual chest CT scan will be performed for current smokers & for those who have quit smoking less than 15 years ago.
  Any patient with a normal PE but positive HPV16 ct-DNA test during follow-up period will require a confirmation test ~1-2 months later.
  If HPV16 ct-DNA positivity is confirmed, an H&N MRI /PET-CT will be performed. Then:
  * If MRI and PET-CT are negative, the patient will be examined every 2 months (PE and HPV16 Ct-DNA dosing) and MRI/PET-CT will be repeated every 4-6 months, until HPV16 Ct-DNA becomes undetectable.
  * If MRI and/or PET-CT is positive, the patient will get a biopsy to confirm disease recurrence. Once confirmed, the patient will have the necessary care, as per local practices, but will continue to be followed up within this study up to 5 years after treatment.
  Interventions: Biological: HPV16 Ct-DNA dosing

INTERVENTIONS:
Biological: HPV16 Ct-DNA dosing — Droplet based digital PCR (ddPCR) technology is a novel method for performing digital PCR. A sample is fractionated into 20,000 droplets, PCR amplification of the template molecules occurs in each individual droplet.
  ddPCR allows to generate quantitative and accurate data without standard curves and also present higher sensitivity compared to conventional quantitative PCR (qPCR). Indeed, this method is based on the realization of millions of single-molecule PCRs in parallel in independent compartment (here droplets of an emulsion) and consequently avoids the bias seen in conventional PCR.
  ddPCR offers an optimized approach for the sensitive detection and quantification of low-target-abundance biological samples.
  DNA extraction will be planned on 1 mL of plasma, which will further increase the sensitivity of our technique initially based on only 200µL of DNA extracted plasma.
  Arms: Lightened follow-up visits frequency (9 visits over 5 years), with HPV16 Ct-DNA dosing

SUMMARY:
SURVEILLE-HPV - A new post therapeutic surveillance strategy for HPV-driven oropharyngeal cancer based on HPV Circulating DNA measures.

HPV-positive oropharyngeal cancer patients have a much better prognosis that their HPV-negative counterparts. Despite this, Post Treatment Surveillance (PTS) strategy does not take into account HPV status.

HPV Circulating DNA (HPV Ct DNA) has emerged as a promising tool to assess the risk of cancer recurrence following treatment. We assume that this biomarker could be helpful to guide PTS.

The number of systematic PTS visits could be significantly reduced in patients with undetectable HPV Ct DNA whereas a closer clinical and radiological follow up could be performed in case of detectable HPV Ct DNA.

If confirmed, this new strategy could have several benefits including:

* reduction of PTS visits for most HPV-positive patients which implies a potential cost decrease and
* Identification of relapse at early stages (before the occurrence of symptoms)

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or over
2. Patient with p16 positive Oropharyngeal squamous cell carcinoma (OPSCC)
3. Clinical stage T1-4, N0-3, M0 (stages I-III)
4. Any tobacco status
5. Life expectancy greater than 36 months
6. Positive HPV16 Ct-DNA measured before curative anticancer treatment
7. Treated by any curative treatment
8. Complete response at 3 months after end of treatment, which means:

   * Undetectable HPV16 Ct-DNA and no residual disease on imaging (group A) or
   * Undetectable HPV16 Ct-DNA and suspicious imaging but persistent disease excluded by either biopsy or repeated imaging (group B1) or
   * Positive HPV16 Ct-DNA and no residual disease on imaging but negative HPV16 Ct-DNA on the subsequent assessment. This second test will be done 1-2 months after the first one (group C1).
9. Patient must be affiliated to a Social Security System (or equivalent)
10. Patients must have signed a written informed consent form prior to any trial specific procedures. If the patient is physically unable to give his/her written consent, a trusted person of his/her choice, note related to the investigator or the sponsor, can confirm in writing the patient's consent.

Exclusion Criteria:

1. Uncontrolled intercurrent illness that would limit compliance with study requirements.
2. Active invasive malignancy within 3 years of inclusion except for non-invasive malignancies such as non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured.
3. Any other HPV induced cancer within 5 years
4. Any condition that may jeopardize the patient participation as well as non-contraception for male and female with child-bearing potential, pregnancy or breast-feeding
5. Patient unwilling or unable to comply with the study protocol and follow-up schedule.
6. Participation in another clinical trial with an investigational medical product during the last 30 days prior to the inclusion and during the present study (except if patient is included in the control arm, with placebo or with a product that have a marketed authorization, used as per the summary of product characteristics (SmPC) for the given indication).
7. Patient deprived of liberty or placed under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) of HPV16 ct-DNA | 24 months
  The presence of HPV16 ct-DNA will be evaluated by ddPCR. NPV will be defined as 2 successive HPV16 ct-DNA negative results.

SECONDARY OUTCOMES:
5- year Negative Predictive Value | 48 and 60 months
  The presence of HPV16 ct-DNA will be evaluated by ddPCR. NPV will be defined as 2 successive HPV16 ct-DNA negative results.
Positive Predictive Value (PPV) of HPV16 ct-DNA | 18, 24, 48, and 60 months
  The presence of HPV16 ct-DNA will be evaluated by ddPCR. PPV will be defined as 2 successive HPV16 ct-DNA positive results.
Rate of relapses detected by HPV16 ct-DNA | 5.5 years
  The proportion of patients with relapse detected by HPV16 ct-DNA without any other symptoms.
Disease-free survival | 5.5 years
  Disease-free survival (DFS) is defined as the delay between date of inclusion and tumor relapse (local, regional, or distant) or death from any cause, whichever occurs first.
Loco-Regional recurrence | From randomization to disease recurrence, up to 5.5 years
  Evaluation of the stage of the first loco-regional event detected by medical imaging. The stage will be defined by the size of the tumor and the number of invaded lymph nodes.
Time of distant recurrence | From randomization to disease recurrence, up to 5.5 years
  The length of time until manifestation of the first metastatic event detected by medical imaging.
Overall survival | From randomization to death from any cause, up to 5.5 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Cost-effectiveness analysis of the proposed strategy | 5.5 years
  To evaluate the economic cost of the lightened surveillance as compared to the standard treatment in terms of cost assessments and incremental cost-effectiveness ratio.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Clinique St Vincent- Réunion, Saint-Denis, La Réunion
  - ISC Avignon, Avignon
  - Georges-François Leclerc, Dijon
  - Oscar Lambret- Lille, Lille
  - La Timone-AP-HM Marseille, Marseille
  - Antoine Lacassagne - NICE, Nice
  - CHU De Nîmes ICG, Nîmes
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Curie - Paris, Paris
  - TENON - APHP Paris, Paris
  - Eugène Marquis-Rennes, Rennes
  - ICO - Site St Herblain, Saint-Herblain
  - ICANS Strasbourg, Strasbourg
  - IUCT Oncopole Toulouse, Toulouse
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided